CLINICAL TRIAL: NCT05659953
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Multiple Ascending Dose and Food Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LMT503 in Healthy Subjects
Brief Title: LMT503 First-in-human SAD, MAD, and FE Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lmito Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMT503-101
Record Dates: First submitted 2022-11-25; First posted 2022-12-21 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Disease; Colitis, Ulcerative; Crohn Disease
Keywords: Macrophage Polarization; Cell metabolism modulation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMT503 (Experimental): Subjects receiving LMT503 orally
  Interventions: Drug: LMT503
- Placebo (Placebo Comparator): Subjects receiving Matched Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LMT503 — Subjects will receive one of several different oral doses of LMT503 once daily
  Arms: LMT503
Drug: Placebo — Subjects will receive one of several different oral doses of Placebo once daily
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled study, consisting of a single ascending dose (SAD) part with integrated food effect (FE) arm, and a multiple ascending dose (MAD) part to assess the safety, tolerability, and PK of ascending single and multiple oral doses of LMT503. The study will start with the SAD part.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 65 years, inclusive, at screening
* Weight : 50 to 110 kg, inclusive, at screening
* Body mass index : 18.0 to 30.0 kg/m2, inclusive, at screening
* At screening, females can be of childbearing potential (but not pregnant or lactating), or of nonchildbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year postmenopausal [amenorrhea duration of 12 consecutive months]); nonpregnancy will be confirmed for all females by a negative serum pregnancy test at screening, (each) admission, and follow-up.
* Female subjects of childbearing potential who have a fertile male sexual partner must agree to use adequate contraception from at least 4 weeks prior to (first) administration of the study drug until 90 days after the follow up visit. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, a cervical cap, or a condom. Total abstinence from heterosexual intercourse, in accordance with the lifestyle of the subject, is also acceptable.
* Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from (first) admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner, if she is of childbearing potential) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, a cervical cap, or a condom. Total abstinence from heterosexual intercourse, in accordance with the lifestyle of the subject, is also acceptable.
* Supine systolic blood pressure between 90 to 140 mmHg, inclusive, diastolic blood pressure between 45 to 90 mmHg, inclusive, and a heart rate between 40 to 100 bpm, inclusive, at screening. If initial results do not meet these criteria, blood pressure may be repeated if in the judgment of the Investigator there is a reason to believe the initial result is inaccurate.
* All prescribed medication must have been stopped at least 30 days prior to (first) admission to the clinical research center. An exception is made for hormonal contraceptives, which may be used throughout the study.
* All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's wort) must have been stopped at least 14 days prior to (first) admission to the clinical research center. An exception is made for paracetamol, which is allowed up to admission to the clinical research center.
* Ability and willingness to abstain from alcohol from 48 hours (2 days) prior to screening and (first) admission to the clinical research center.
* Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) and grapefruit (juice) from 48 hours (2 days) prior to (each) admission to the clinical research center.
* Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
* Willing and able to sign the ICF.

Exclusion Criteria:

* Previous participation in the current study.
* Employee of ICON or the Sponsor.
* History of relevant drug and/or food allergies.
* Using tobacco products within 2 months prior to (first) admission.
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
* Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, gamma hydroxybutyric acid, tricyclic antidepressants, and alcohol) at screening or (at one of the) admission(s) to the clinical research center.
* Average intake of more than 24 units of alcohol per week: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits).
* Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) 1 and 2 antibodies.
* Participation in a drug study within 30 days prior to (the first) drug administration in the current study. Participation in 4 or more other drug studies in the 12 months prior to (the first) drug administration in the current study.
* Donation or loss of more than 450 mL of blood within 60 days prior to (the first) drug administration. Donation or loss of more than 1.5 liters of blood (for male subjects)/more than 1.0 liters of blood (for female subjects) in the 10 months prior to (the first) drug administration in the current study.
* Significant and/or acute illness within 5 days prior to (the first) drug administration that may impact safety assessments, in the opinion of the Investigator.
* Unwillingness to consume the FDA breakfast.
* Unsuitable veins for infusion or blood sampling.
* Vaccination against SARS-CoV-2 planned between 2 weeks prior to (first) admission and follow-up.
* Positive nasopharyngeal PCR test for SARS-CoV-2 on Day -1 or if there was any known close contact with a person who tested positive for SARS-CoV-2 or with a COVID-19 patient within 2 weeks prior to admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) in the SAD and MAD part | up to Day 17
  Incidence and severity of AEs including clinical significant changes in safety laboratory, vital signs, 12-lead ECG, continuous cardiac monitoring (telemetry), and physical examination

SECONDARY OUTCOMES:
PK parameter | up to Day 10, 72 hours post dose
  Maximum observed concentration (Cmax) of LMT503 in plasma
PK parameter | up to Day 10, 72 hours post dose
  Time to maximum observed concentration (Tmax) of LMT503 in plasma
PK parameter | up to Day 10, 72 hours post dose
  Apparent terminal elimination half-life (t1/2) of LMT503 in plasma
PK parameter | up to Day 10, 72 hours post dose
  Area under the plasma concentration-time curve from time 0 to time tau (AUC0-tau) of LMT503 in plasma
PK parameter | up to Day 10, 72 hours post dose
  Terminal elimination rate constant (kel) of LMT503 in plasma
PK parameter | up to Day 10, 72 hours post dose
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of LMT503 in plasma (SAD and FE part)
PK parameter | up to Day 10, 72 hours post dose
  Area under the plasma concentration-time curve up to time t (AUC0-t) of LMT503 in plasma (SAD and FE part)
PK parameter | up to Day 10, 72 hours post dose
  Concentration at the end of the dosing interval (Ctrough) of LMT503 in plasma (MAD only)
PK parameter | up to Day 10, 72 hours post dose
  Cumulative amount of LMT503 excreted in urine to time t (Aeurine) (SAD and FE part)
PK parameter | up to Day 10, 72 hours post dose
  Cumulative amount of LMT503 excreted in urine to time tau (Aeurine,ss) (MAD only)
Number of Treatment Emergent Adverse Events (TEAEs) in Food Effect part | up to Day 4, 72 hours post dose
  Incidence and severity of AEs including clinical significant changes in safety laboratory, vital signs, 12-lead ECG, continuous cardiac monitoring (telemetry), and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Wheeseong LEE, PhD, Study Chair — Lmito Therapeutics Inc.
Locations (1):
- ICON plc Company - Early Development Services, Groningen, NZ, Netherlands

IPD SHARING:
Plan to Share IPD: No